CLINICAL TRIAL: NCT07329712
Title: Comparing Tear Proteomics Profile in Dry Eye Disease pre-and Post-treatment With Low Level Light Therapy
Status: Recruiting | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Other Study IDs: 2025-0870; 2025-0870 (Other: Singhealth CIRB)
Record Dates: First submitted 2025-12-21; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction (Disorder)
Keywords: Dry Eye; low level light therapy; Eyelight; Tears proteomics; tear cytokine; MGD
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tears Sample (Schirmers Test)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing low level light therapy

SUMMARY:
The purpose of this research study is to understand the mechanism of action of low level light therapy and also potentially yield markers associated with good treatment response. Low-level light therapy is light-based treatment delivered through advance eye-light device. This therapy uses light energy to provide energy to the meibomian gland cells to slow down age-ing, improve tear stability and reduce inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Must be eligible for, and have consented for low level light therapy
2. Must not have presented to the clinic for an acute eye problem such as visual loss or painful eye
3. Ability to give informed consent.
4. Age more or equals to 21 years old.

Exclusion Criteria:

1. Patients who are unable to or decline to give consent.
2. Age less than 21 years old.
3. Patients who presented to the clinic for an acute eye problem such as visual loss or painful eye.
4. Patients not suitable for low level lighttherapy:

   * Pregnant
   * Fitted with pacemakers, metal, electrical, acoustic prosthetics
   * Epilepsy, cardiac rhythm or frequency disorders
   * Fever, thrombophlebitis or acute phlebitis of the legs, large-sized varicose veins, or venous surgery within 2 months
   * Uncontrolled hypertension or severe diabetes
   * Open wounds on eyelid or skin
   * Evolving cancer or hepatitis
   * Blood anticoagulant or coagulation defect

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing low level light therapy that met the study inclusion and exclusion
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparing tear proteomics profile in dry eye disease pre-and post-treatment with low level light therapy | Baseline visit and Post Baseline visit 3 months (+3 weeks).
  Aim 1: Tear proteomic profile of MGD patients with DED pre- and post-treatment with LLLT will be profiled Aim 2: Baseline tear cytokine levels will be measured using the novel Olink 500-plex technology in DED patients with MGD undergoing LLLT

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Insititute, Singapore, Singapore